CLINICAL TRIAL: NCT01953887
Title: An Open-label, Randomized, Three-period Crossover, Single Dose Study to Compare the Pharmacokinetics of the Final EC905 Formulation to Marketed Solifenacin (Vesicare®) and Tamsulosin OCAS (Omnic OCAS®)
Brief Title: A Study to Compare the Amount of Drug in the Blood After a Single Tablet EC905 Containing Solifenacin and Tamsulosin is Taken by Healthy Males Compared to Separate Tablets of Solifenacin and Tamsulosin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 905-CL-072; 2009-015618-22 (EudraCT Number)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: EC905; Pharmacokinetics; Healthy Subjects
Keywords: Phase I; Final formulation EC905; Solifenacin succinate; Tamsulosin HCl; Marketed drugs
MeSH Terms: interventions — Solifenacin Succinate; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 combination tablet EC905 (Experimental)
  Interventions: Drug: EC905
- 2: solifenacin (Experimental)
  Interventions: Drug: solifenacin
- 3: tamsulosin (Experimental)
  Interventions: Drug: tamsulosin

INTERVENTIONS:
Drug: EC905 — Oral
  Arms: 1 combination tablet EC905
Drug: solifenacin — oral
  Other Names: Vesicare®
  Arms: 2: solifenacin
Drug: tamsulosin — oral
  Other Names: Omnic OCAS®
  Arms: 3: tamsulosin

SUMMARY:
A study to assess the amount of drug in the blood of young to middle aged, healthy, male subjects after they received the final formulation of EC905 compared to solifenacin (Vesicare®) and tamsulosin OCAS (Omnic OCAS®).

Subjects are given a single dose of the combination tablet EC905, Vesicare® and Omnic OCAS® in 3 separate periods.

DETAILED DESCRIPTION:
The subjects are randomized to one of 6 treatment sequence groups.

Subjects are admitted to the clinical unit on Day -1 for pre-dose assessments. They remain in the clinic for two periods of 11 days and one period of 14 days.

After randomization the subjects receive a single dose treatment on Day 1 followed by blood sampling for pharmacokinetic (PK) assessment. For both EC905 and Vesicare®, blood sampling continues for 10 days after dosing; for Omnic OCAS®, it continues for 3 days after dosing.

Each period is separated by a wash-out period of at least 4 day, and subjects are checked for eligibility again one day prior to the start of a new dosing day.

Vital signs, safety ECG measurements, safety laboratory assessments, adverse events and concomitant medications are monitored throughout the investigational period.

A blood sample is drawn for CYP2D6 genotyping, in order to evaluate the effect of the CYP2D6 genotype on the PK of tamsulosin.

Subjects return for an End of Study Visit (ESV) 7 days after the last on-site period, or after withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 18.5 and 30.0 kg/m2, inclusive

Exclusion Criteria:

* Known or suspected hypersensitivity to solifenacin, tamsulosin, EC905, Vesicare, Omnic OCAS or any of the components of the formulations used.
* Any of the contraindications or precautions for use as mentioned in the applicable sections of the SPC's of tamsulosin or solifenacin.
* Use of grapefruit (more than 3 x 200 ml) or marmalade (more than three times) in the week prior to admission to the Clinical Unit, as reported by the subject.
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The Pharmacokinetics (PK) of solifenacin after a single dose of the final formulation of the combination tablet EC905 with a single dose of Vesicare® and Omnic OCAS® | Predose to Day 10 after dosing (22 times)
  AUClast (Area under the curve until last sample taken), Cmax (Maximum concentration)
The Pharmacokinetics (PK) of tamsulosin HCl after a single dose of the final formulation of the combination tablet EC905 with a single dose of Vesicare® and Omnic OCAS® | Predose to Day 10 after dosing (22 times)
  AUClast (Area under the curve until last sample taken), Cmax (Maximum concentration)

SECONDARY OUTCOMES:
The PK of solifenacin and tamsulosin HCl after a single dose of the final formulation of the combination tablet EC905 with a single dose of Vesicare® and Omnic OCAS® | Predose to Day 10 after dosing (22 times)
  AUCinf (AUC extrapolated until infinity), t1/2 (Apparent terminal elimination half-life), tmax (Time to attain Cmax), CL/F (Apparent total body plasma clearance), Vz/F (Apparent volume of distribution)
Safety and tolerability of single doses of the final formulation combined EC905, marketed Vesicare® and marketed Omnic OCAS® | Screening to End of Study Visit (at least 7 days after the last on site period (treatment and PK sampling), or after withdrawal.)
  Adverse events, clinical laboratory tests, vital signs, Electrocardiogram (ECG), physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- Parexel, London, United Kingdom